CLINICAL TRIAL: NCT04243460
Title: Influence of Soft Tissue Thickness on the Marginal Bone Level Around Implants in Esthetic Zone: 1 Year Randomized Control Trail
Brief Title: Influence of Soft Tissue Thickness on the Bone Level Around Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Innovation Center Wroclaw (Other)
Collaborators: Camlog Oral Reconstruction Foundation (Other); Wrocław Medical University (Unknown)
Responsible Party: Principal Investigator, Jakub Hadzik, DDS, PhD, Principal Investigator, Medical Innovation Center Wroclaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STT and MBL
Record Dates: First submitted 2020-01-11; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Tooth Loss
Keywords: Dental Implants
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTG connective tissue graft augmentation (Experimental): CTG connective tissue graft (CTG) was used for soft tissue augmentation. I
  Interventions: Procedure: Connective tissue graft augmentation (CTG)
- XCM Xenogeneic collagen matrix (XCM)graft augmentation (Active Comparator): Xenogeneic collagen matrix (XCM) was used for soft tissue augmentation.
  Interventions: Procedure: Xenogeneic collagen matrix (XCM) graft augmentation

INTERVENTIONS:
Procedure: Xenogeneic collagen matrix (XCM) graft augmentation — 12 months after gingival augmentation Measurement of marginal bone level and soft tissue thickness were done. STT (soft tissue thickness) was measured using ultrasonography with a Pirop® dental, ultrasound device (Echoson Company, Poland). The patients underwent a clinical and ultrasound examination before, 3 and 12 months after gingival augmentation (GA) respectively to evaluate TKT at two points using ultrasound equipment (Pirop®, Echoson).
  Intraoral radiographs were taken using a paralleling technique with a Rinn-type film holder in high resolution mode (Visualixe HD®, Gendex®, USA). Two images of each region were selected to calculate the marginal bone changes:
  Arms: XCM Xenogeneic collagen matrix (XCM)graft augmentation
Procedure: Connective tissue graft augmentation (CTG) — 12 months after gingival augmentation Measurement of marginal bone level and soft tissue thickness were done. STT (soft tissue thickness) was measured using ultrasonography with a Pirop® dental, ultrasound device (Echoson Company, Poland). The patients underwent a clinical and ultrasound examination before, 3 and 12 months after gingival augmentation (GA) respectively to evaluate STT (soft tissue thickness) at two points using ultrasound equipment (Pirop®, Echoson).
  Arms: CTG connective tissue graft augmentation

SUMMARY:
Healthy soft tissue around the implant are considered as a biological seal to prevent inflammatory periimplant diseases and ensure healthy, stable and long-term survival of a dental implant. Due to the fact that the measurement methods in the literature differ, it is necessary to establish objective measurement method and to determine the minimum amount of tissue thickness to maintain a stable level of bone around the implant.

DETAILED DESCRIPTION:
Healthy soft tissue around the implant are considered as a biological seal to prevent inflammatory periimplant diseases and ensure healthy, stable and long-term survival of a dental implant. Due to the fact that the measurement methods in the literature differ, it is necessary to establish objective measurement method and to determine the minimum amount of tissue thickness to maintain a stable level of bone around the implant.

Purpose:

The aim of the study was to determine the effect of soft tissues in the implant area on the marginal bone level loss in the implant area and to define of the critical gingival thickness to minimize marginal bone level (MBL) loss.

Materials and methods:

75 bone level implants (Conelog® Camlog, Switzerland) were inserted in the aesthetic area. Thickening of soft tissues was performed both before and after implantation (group II and III), CTG and XCM were used (subgroup a and b). 12 months after the loading with final restoration, the thickness of soft tissues in the implant area was examined with ultrasonography (USG) device (Pirop®, Echoson, Poland), and each implant was subjected to Radiovisiography (RVG) RVG examination, where MBL loss was determined.

ELIGIBILITY:
Inclusion Criteria:

To qualify for the study, the patients had to be >18 years and have missing teeth in the esthetic zone. Additional inclusion criteria were as follows:

* missing single or double teeth in the anterior area of their upper or lower jaw with a proper inter arch relationship (incisors, canines and first premolar) with a ridge width (bucco-lingual) greater than 5 mm at its narrowest point and a minimum keratinized gingiva height of 2 mm buccally.
* No previous soft tissue augmentation procedure at experimental site

Exclusion Criteria:

The criteria that disqualified patients from the study were previous grafting procedures in the area of interest and systemic or local diseases that could compromise healing or osteointegration. Smokers and patients with bruxism were also excluded from the study. Additional exclusion criteria were as follows:

* implants placed with an insertion torque of 35 Ncm or less;
* irradiation in the head and neck area;
* untreated periodontitis;
* poor oral hygiene (plaque score Approximal Plaque Index (API) 20%, bleeding score 10%) and
* poor motivation;
* fresh post extraction sockets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound examination | 12 months
  ultrasound USG examination of tissue hickness
Radiological examination | 12 monhs
  RVG examination of marginal bone level change

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Hadzik, PhD, DDS, Principal Investigator — jakub.hadzik@umed.wroc.pl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puzio M, Blaszczyszyn A, Hadzik J, Dominiak M. Ultrasound assessment of soft tissue augmentation around implants in the aesthetic zone using a connective tissue graft and xenogeneic collagen matrix - 1-year randomised follow-up. Ann Anat. 2018 May;217:129-141. doi: 10.1016/j.aanat.2017.11.003. Epub 2017 Dec 15. PMID 29248711